CLINICAL TRIAL: NCT02693925
Title: Sleep-related Breathing Disorders in Cardiological Outpatients From a German University Clinic - Prevalence, Classification, Diagnostic Accuracy
Brief Title: Sleep-related Breathing Disorders in Cardiological Outpatients
Acronym: SRBD-Cardio
Status: Completed | Type: Observational
Sponsor: Wissenschaftliches Institut Bethanien e.V (Other)
Collaborators: University Clinic Cologne (Unknown)
Responsible Party: Sponsor
Other Study IDs: WI_SBASKardio_14-322
Record Dates: First submitted 2016-02-17; First posted 2016-02-29 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the prevalence of sleep-related breathing disorders (SRBD) in clinically stable cardiologic outpatients of a German university clinic by means of polygraphy.

Furthermore, the practicability of the underlying diagnostic process in clinical application is assessed as well as the sensitivity and specificity of polygraphy as compared to the reference standard of polysomnography. Another aim is to determine the individual cardiovascular risk profile by pulse wave analysis and risk classification according to European Society of Hypertension (ESH) and European Society of Cardiology (ESC), "ESH/ESC risk".

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Present chronic cardiovascular disease (incl. but not limited to: ischemic heart disease, arterial hypertension, heart failure, atrial fibrillation)
* Current clinically stable state (incl. patients after a cardiovascular-related, emergency hospital admission and subsequent recompensation towards the end of their hospital stay

Exclusion Criteria:

* Age <18 years
* Acute life-threatening disease (incl. but not limited to:instable angina pectoris, acute bronchial asthma, heart failure New York Heart Association (NYHA) stage IV, myocardial infarction, exacerbated chronic obstructive pulmonary disease (COPD), Malignant disease requiring treatment)
* Pregnancy and/or lactation
* Any medical, psychological or other condition impairing the patient's ability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cardiologic diseases who have a routine outpatient follow-up visit in the heart center of the University Clinic Cologne or are at the end of a cardivascular-related hospital stay in stable (recompensated) state.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-12-16 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Prevalence of sleep-related breathing disorders | Once within two days of inclusion
  Prevalence of sleep-related breathing disorders as measured by ambulatory polygraphy and defined as an respiratory disturbance index of >=15/h

SECONDARY OUTCOMES:
Number of patients included | through study completion, an average of 21 months
  Total number of patients included in the study after overall study conclusion
Number of patients with actually performed polygraphy | through study completion, an average of 21 months
  Total number of patients in whom ambulatory polygraphy was actually performed, after overall study conclusion
Number of patients with assessable polygraphy | through study completion, an average of 21 months
  Total number of patients in whom ambulatory polygraphy was assessable, after overall study conclusion
Number of patients with actually performed polysomnography | through study completion, an average of 21 months
  Total number of patients in whom stationary polysomnography was actually performed, after overall study conclusion
Number of patients with assessable polysomnography | through study completion, an average of 21 months
  Total number of patients in whom stationary polysomnography was assessable, after overall study conclusion

CONTACTS AND LOCATIONS:
Overall Officials: Winfried J Randerath, Prof. Dr., Principal Investigator — Wissenschaftliches Institut Bethanien e.V
Locations (1):
- University Clinic Cologne, Heart Center, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No